CLINICAL TRIAL: NCT03033589
Title: Femoral Nerve Block Versus. Adductor Canal Nerve Block for Peri-Operative Analgesia Following Anterior Cruciate Ligament Reconstruction: Evaluation of Post-Operative Pain and Strength
Brief Title: Femoral Nerve Block Versus Adductor Canal Nerve Block for Peri-Operative Analgesia Following Anterior Cruciate Ligament (ACL) Reconstruction: Evaluation of Post-operative Pain and Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Charles S Day, Orthopedic Surgeon, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10083
Record Dates: First submitted 2016-08-24; First posted 2017-01-27 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Pain
Keywords: Pain control; Anterior Cruciate Ligament (ACL_ Reconstruction); Regional Anesthesia
MeSH Terms: conditions — Pain; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adductor Canal Nerve Block (Active Comparator): One hour prior to procedure, subject to receive 20 mL of 0.5% ropivacaine injected into the sheath of the saphenous nerve at the adductor hiatus. Ultrasound guidance utilized for appropriate localization of the targeted nerve sheath for local infiltration. No nerve stimulators to be utilized during or after the procedure.
  Interventions: Drug: Marcaine 0.25 % Injectable Solution
- Femoral Nerve block (Active Comparator): One hour prior to procedure, subject to receive 30 mL of 0.5% ropivacaine injected into the nerve sheath of the femoral nerve at the level of the femoral triangle. Ultrasound guidance utilized for appropriate localization of the targeted nerve sheath for local infiltration. No nerve stimulators to be utilized during or after the procedure.
  Interventions: Drug: Marcaine 0.25 % Injectable Solution

INTERVENTIONS:
Drug: Marcaine 0.25 % Injectable Solution — For the adductor canal block, 20 mL of 0.25% marcaine will be injected with the use of ultrasound guidance into the adductor canal by the attending anesthesiologist on the case in the pre-op holding area.
  Arms: Adductor Canal Nerve Block
Drug: Marcaine 0.25 % Injectable Solution — For the femoral nerve block, 30 mL of 0.25% marcaine will be injected with the use of ultrasound guidance around the femoral nerve sheath by the attending anesthesiologist on the case in the pre-op holding area.
  Arms: Femoral Nerve block

SUMMARY:
All patients over the age of 16 undergoing primary or revision anterior cruciate ligament reconstruction with the use of bone-patellar-bone autograft are eligible for the study. Patients will be randomized pre-operatively to receive either an adductor canal nerve block (single injection) or a femoral nerve block (single injection). Post-operatively, the primary outcome measures of pain level using visual analog scale as well as narcotic and non-narcotic analgesic requirements will be measured.

DETAILED DESCRIPTION:
Currently, because of its good track record, femoral nerve block is the modality of choice for post-operative pain control following elective anterior cruciate ligament reconstruction at our institution. It has been proven in the literature to provide good post-operative pain analgesia following this procedure (1). However, femoral nerve block is not without its concerns, including the concern for long-term quadriceps weakness (2). Benefits of decreased use of Femoral Nerve Block include the decreased incidence of side effects and/or complications, and use of quadriceps for immediate rehabilitation. Benefits of Adductor canal nerve block include possible equivalent pain control with the avoidance of motor de-innervation and its deleterious adverse effect of quadriceps weakness postoperatively. Adductor canal nerve block has proven to be effective in other orthopaedic procedures involving the knee including total knee arthroplasty (3). This results of this study will give more information on how to better control pain in the post-op period while minimizing the deleterious side effects for patients undergoing ACLreconstruction.

All patients over the age of 16 undergoing primary or revision anterior cruciate ligament reconstruction with the use of bone-patellar-bone autograft are eligible for the study. Patients will be randomized pre-operatively to receive either an adductor canal nerve block (single injection) or a femoral nerve block (single injection). A single dose of 30 mL of 0.25% marcaine is injected for femoral nerve block and 20 mL of 0.25% marcaine for Adductor Canal nerve block. These procedures will be performed by the attending anesthesiologist prior to surgery. After surgery the patient will record their pain levels using visual analog scale (VAS) score in a daily diary for the first 5 post-operative days. They will also record all medication requirements, both narcotic and non-narcotic analgesic medications. The patient will be tested on their ability to perform a straight leg raise in the post-anesthesia care unit (PACU) and at their first post-operative visit.

ELIGIBILITY:
Inclusion Criteria:

* Primary ACL Reconstruction with use of Bone-Patellar-Bone Autograft
* Age 16 or older

Exclusion Criteria:

* Patients under 16
* The use of Allograft,
* The use of hamstring autograft
* The use quadriceps autograft
* Patients allergic to active ingredients in the injection.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Post-op Day 0-5
  Every 4 hours the patient will record in their study binder their pain level on a scale from 1-10. They are instructed that a 1 signifies minimal pain that is nearly unnoticeable whereas a pain scale of 10 is the most intolerable pain imaginable.
Narcotic Requirement | Post-op Day 0-5
  Every time a the prescribed narcotic is consumed, in this study it is Norco 5-325 (Hydrocodone-Acetaminophen), the subject is instructed to log their quantity consumed as well as the time consumed in the study binder provided to them

SECONDARY OUTCOMES:
Thigh circumference | 2 weeks post-operative vs 6 months post-operative
  Thigh circumference will be measured 10 cm above the superior pole of the patella for both the operative and non-operative thighs.
Straight Leg Raise | 0-7 days post-operative
  We will test the ability to perform straight leg raise in post-anesthesia care unit as well as at first post-operative visit (5-7 days post-operative).

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System - CFP 642, Detroit, Michigan, United States

REFERENCES:
- [Background] Guirro UB, Tambara EM, Munhoz FR. Femoral nerve block: Assessment of postoperative analgesia in arthroscopic anterior cruciate ligament reconstruction. Braz J Anesthesiol. 2013 Nov-Dec;63(6):483-91. doi: 10.1016/j.bjane.2013.09.001. Epub 2013 Dec 5. PMID 24565346
- [Background] Luo TD, Ashraf A, Dahm DL, Stuart MJ, McIntosh AL. Femoral nerve block is associated with persistent strength deficits at 6 months after anterior cruciate ligament reconstruction in pediatric and adolescent patients. Am J Sports Med. 2015 Feb;43(2):331-6. doi: 10.1177/0363546514559823. Epub 2014 Dec 2. PMID 25466410
- [Background] Kim DH, Lin Y, Goytizolo EA, Kahn RL, Maalouf DB, Manohar A, Patt ML, Goon AK, Lee YY, Ma Y, Yadeau JT. Adductor canal block versus femoral nerve block for total knee arthroplasty: a prospective, randomized, controlled trial. Anesthesiology. 2014 Mar;120(3):540-50. doi: 10.1097/ALN.0000000000000119. PMID 24401769
- [Derived] Lynch JR, Okoroha KR, Lizzio V, Yu CC, Jildeh TR, Moutzouros V. Adductor Canal Block Versus Femoral Nerve Block for Pain Control After Anterior Cruciate Ligament Reconstruction: A Prospective Randomized Trial. Am J Sports Med. 2019 Feb;47(2):355-363. doi: 10.1177/0363546518815874. Epub 2018 Dec 17. PMID 30557034